CLINICAL TRIAL: NCT05748860
Title: PRecision Ecmo in CardIogenic Shock Evaluation
Acronym: PRECISE
Status: Not yet recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/AB003
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cardiogenic Shock
Keywords: ECMO; cardiogenic shock; ECPR; critical illness; intensive care
MeSH Terms: conditions — Shock, Cardiogenic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biomarkers of interest for the PRECISE Study include biomarkers involved in neuroprognositication (neuron specific enolase, neurofilament), mortality prediction (lactate), heart failure (Troponin, pro BNP), endothelial damage (Angiopoietin 2), inflammation and other biomarkers that may be involved in risk prediction. We will also collect samples of free genetic material (eg free mitochondria), which will not involve genome wide association, and therefore will not include information about heritable diseases in families.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients commencing on VA-ECMO: The study population is adult patients on VA-ECMO for cardiogenic shock or cardiac arrest that are or will be enrolled in the national ECMO registry (EXCEL).

SUMMARY:
Venoarterial (VA) ECMO is a form of life support for patients with severe cardiogenic shock and cardiac arrest. Although it can be lifesaving, currently many patients still die or have long term disability, such as weakness, shortness of breath and cognitive impairments, and it remains extremely expensive. It is important that new ways of identifying which patients will gain the most benefit from ECMO are found, while also avoiding costly futile use when it there is no benefit.

The PRECISE Study is an Australian-led, nation-wide observational study that will investigate whether biomarkers can better guide decisions around to whom and how ECMO is delivered. The study will involve the collection of a small amount of blood (which would normally be discarded) at up to 4 different time points, including just prior to ECMO initiation, and also at days 1, 3, and 7 of ECMO support. These results will then be linked to a national registry which includes the important patient centred outcomes, such as disability at 6 months. This study will lead to the better support of a highly vulnerable population, and improve the efficiency of one of the most complex and costly interventions available.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be commencing on VA ECMO (for cardiogenic shock or ECPR)
* 18 years old or older
* Patients who will be enrolled in the EXCEL Registry (HREC Project 534/18)

Exclusion Criteria:

* Patients who are already on ECMO, or where
* There are inadequate resources to complete the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is adult patients on VA-ECMO for cardiogenic shock or cardiac arrest that are or will be enrolled in the national ECMO registry (EXCEL: HREC Project 534/18).
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability-free survival at day 180 | Day 180
  Measured with the World Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Aidan JC Burrell, Principal Investigator — Australian and New Zealand Intensive Care Research Centre

IPD SHARING:
Plan to Share IPD: Undecided